CLINICAL TRIAL: NCT05127460
Title: Computer-assisted Atrial Fibrillation Risk Detection In Oral-anticoagulant Use, Lowering Stroke Risk, and Optimizing Guidance With an Intelligent Screening Tool (CARDIOLOGIST): a Pragmatic Randomized Controlled Trial
Brief Title: CARDIOLOGIST Trial: Artificial Intelligence Enabled Electrocardiogram for Atrial Fibrillation Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2021002
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation New Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will have access to the screening tool.
  Interventions: Other: AI-enabled ECG-based Screening Tool
- Control (No Intervention): Patients randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool — Primary care clinicians in the intervention group had access to the report, which displayed whether the AI-ECG result was positive or negative. The system will send a message to corresponding physicians if positive finding.
  Arms: Intervention

SUMMARY:
This is a randomized controlled trial (RCT) to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis and management of Atrial Fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in emergency department or inpatient department
* Patients had at least 1 ECG
* Patients cared by non-cardiologist

Exclusion Criteria:

* Patients without history of atrial fibrillation diagnosis.
* Patients without history of long-term NOAC or warfarin usage.
* Patients without history of hemorrhagic stoke or ishemic stroke.
* Patients with low eGFR (<30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25732 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of taking AF treatment medications | Within 90 days
  defined as use of long-term NOAC (apixaban, rivaroxaban, endoxaban, dabigatran).
Proportion of ischemic Stroke | Within 90 days
  After performing an electrocardiogram, the patient's physical conditions is tracked.

SECONDARY OUTCOMES:
Proportion of cardiologist consultation | Within 90 days
  Cardiovascular outpatient visit after discovering atrial fibrillation.
Proportion of new-onset AF diagnosis | Within 90 days
  Atrial fibrillation diagnosis in medical records
Proportion of echocardiogram performed after ECGs | Within 90 days
  After performing the ECG examination, perform the echocardiography examination.
Proportion of new-onset heart failure | Within 90 days
  After performing an electrocardiogram, the patient's medical record is tracked.
Proportion of gastrointestinal bleeding | Within 90 days
  After performing an electrocardiogram, the patient's medical record is tracked.
Proportion of hemorrhagic stroke | Within 90 days
  After performing an electrocardiogram, the patient's medical record is tracked.
Proportion of all cause mortality(death) | Within 90 days
  After performing an electrocardiogram, the patient's survival is tracked.

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu WT, Lin C, Lee CC, Chang CH, Fang WH, Tsai DJ, Lin WY, Hung Y, Chen KC, Lee CH, Tsai TN, Lin WS, Hung YJ, Lin SH, Tsai CS, Lin CS. Artificial Intelligence-Enabled ECGs for Atrial Fibrillation Identification and Enhanced Oral Anticoagulant Adoption: A Pragmatic Randomized Clinical Trial. J Am Heart Assoc. 2025 Jul 15;14(14):e042106. doi: 10.1161/JAHA.125.042106. Epub 2025 Jul 3. PMID 40611485